CLINICAL TRIAL: NCT03427658
Title: Impact of Repeated Sweet and Non-sweet Food Consumption on Subsequent Sweet Food Preferences and Intake
Brief Title: Repeated Sweet Consumption and Subsequent Sweet Food Preferences and Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bournemouth University (Other)
Collaborators: University of Bristol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PRKA2018
Record Dates: First submitted 2018-02-01; First posted 2018-02-09 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-01

CONDITIONS: Repeated Sweet Food Consumption
Keywords: sweet taste; food preferences; food intake
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Intervention allocation will be undertaken by a researcher not in direct contact with any one participant, following randomization by drawing lots.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increase sweet food consumption (Experimental): Participants are asked to increase their consumption of sweet foods throughout their diet. Participants will be supported through an individual dietary interview where sweet foods will be highlighted and additional sweet food consumption recommended.
  Interventions: Behavioral: Sweet food consumption
- Decrease sweet food consumption (Active Comparator): Participants are asked to decrease their consumption of sweet foods throughout their diet. Participants will be supported through an individual dietary interview where sweet foods will be highlighted and substitutions for sweet food consumption will be recommended.
  Interventions: Behavioral: Sweet food consumption

INTERVENTIONS:
Behavioral: Sweet food consumption — Comparison of the impacts of sweet and non-sweet food consumption

SUMMARY:
This study will assess the impact of repeated sweet versus non-sweet food consumption on subsequent sweet and non-sweet food preferences and intakes

DETAILED DESCRIPTION:
Participants will be randomized to receive instructions to either increase or decrease sweet food consumption for 6 days, and impacts on food preferences and intakes will be assessed at baseline and after 1 week. Preferences for sweet and non-sweet foods will be assessed during two taste tests at each assessment time, where six different foods will be rated. Sweet and non-sweet food consumption will also be measured at two meals at each assessment time - breakfast and lunch. Identical buffet meals composed of sweet and non-sweet foods suitable for consumption at breakfast and lunch will be provided ad-libitum.

ELIGIBILITY:
Inclusion Criteria:

* No known food allergy
* No known taste or appetite allergies
* Non-smokers
* Do not habitually consume exclusively / almost exclusively a sweet or non-sweet diet
* Able to provide consent and complete all study measures

Race / ethnicity will not be requested.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rogers, PhD, Principal Investigator — University of Bristol; Katherine Appleton, PhD, Principal Investigator — Bournemouth University, UK
Locations (1):
- University of Bristol, Bristol, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol is currently available from the PI on reasonable request. All generated data will be available from the PI, following completion and publication of the work on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following completion and publication of the study. Data will be stored for ten years following publication of the work.
Access Criteria: Direct contact and reasonable request of the PI

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption
Started | 21 | 15
Completed | 21 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption | Total
Number analyzed (Participants) | 21 | 15 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.0 (1.0) | 21.3 (0.8) | 21.1 (0.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 6 | 6 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 21 | 15 | 36

OUTCOME MEASURES:

1. Primary Outcome: Food Preferences
Description: Ratings of three sweet and three non-sweet foods during a taste test (two tests). Measures are made on a visual analogue scale from 0 (not at all) to 100 (extremely), where higher scores denote higher preferences.
Time Frame: Change from Baseline to 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption
Number analyzed (Participants) | 21 | 15
units on a scale | 7 (19) | 1 (13)

2. Primary Outcome: Food Intake
Description: Amount of sweet and non-sweet foods consumed during breakfast and lunch. Measures are made of grams of each sweet food consumed.
Time Frame: Change from Baseline to 1 week
Measure: Mean (Standard Deviation); unit: grams sweet food
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption
Number analyzed (Participants) | 21 | 15
grams sweet food | -24 (189) | -15 (183)

3. Secondary Outcome: Hunger Ratings
Description: Ratings of subjective perceptions (two meals). Measures are made on a visual analogue scale from 0 (not at all) to 100 (extremely), where higher scores denote higher hunger.
Time Frame: Change from Baseline to 1 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption
Number analyzed (Participants) | 21 | 15
units on a scale | 7 (28) | -2 (35)

ADVERSE EVENTS:
Time Frame: 1 week
Description: All participants are asked if they experienced any difficulties. Adverse events are disclosed voluntarily and spontaneously by participants.
Arm/Group | Increase Sweet Food Consumption | Decrease Sweet Food Consumption
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/15
Other Adverse Events (participants affected / at risk) | 0/21 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03427658/Prot_SAP_000.pdf